CLINICAL TRIAL: NCT00494325
Title: The Role of Macular Pigment in Patients With Age-related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Sebastian Wolf, Director, Insel Gruppe AG, University Hospital Bern
Other Study IDs: KEK 73/05; SNF 3200 Bo-109962/1 (Other Grant/Funding Number: SNF)
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Age Related Maculopathy
Keywords: age related maculopathy, macular pigment
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In the industrialised world age-related macular degeneration (ARMD) is the leading cause for legal blindness beyond the age of 50 years. Recent studies indicate that the amount and status of the macular pigment (MP) may play a central role in the development and progression of the disease. It has been demonstrated that the MP density can be increased by dietary supplementation. First results of MP density measurements with a modified confocal laser scanning ophthalmoscope show that this method allows to quantify the MP in a clinical setting. The aim of this study is to assess the peak MP density as well as the MP distribution in relation to the risk for ARMD. We will establish reference values for MP density distribution in a normal population and compare these to values obtained from patients with age related maculopathy in a cross-sectional study. For all MP density measurements we will use a modified scanning laser ophthalmoscope and dietary intake of macular pigment will be assessed using a Food Frequency Questionnaire. Clinical examinations will include ETDRS visual acuity, binocular ophthalmoscopy, colour fundus photography and autofluorescence imaging. The results of our study will help assess the relationship of macular pigment density and distribution with ARMD. Additionally, we will be able to identify patients with low MP density, and probably improve the early diagnosis of patients at high risk for developing ARMD. This will be the basis for dietary supplementation of lutein and/or zeaxanthin in patients with high risk for ARMD due to low macular pigment values.

ELIGIBILITY:
Inclusion Criteria:

* age related maculopathy

Exclusion Criteria:

* other macular diseases

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with early ARM
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2005-10; Primary Completion 2010-12 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of development of late AMD | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Wolf, MD, Principal Investigator — University of Bern; Sebastian Wolf, MD PhD, Study Director — University of Bern
Locations (1):
- Klinik und Poliklinik für Augenheilkunde, University Bern, Bern, Switzerland

REFERENCES:
- [Derived] Wolf-Schnurrbusch UE, Wittwer VV, Ghanem R, Niederhaeuser M, Enzmann V, Framme C, Wolf S. Blue-light versus green-light autofluorescence: lesion size of areas of geographic atrophy. Invest Ophthalmol Vis Sci. 2011 Dec 16;52(13):9497-502. doi: 10.1167/iovs.11-8346. PMID 22110076
- [Derived] Rothenbuehler SP, Wolf-Schnurrbusch UE, Wolf S. Macular pigment density at the site of altered fundus autofluorescence. Graefes Arch Clin Exp Ophthalmol. 2011 Apr;249(4):499-504. doi: 10.1007/s00417-010-1528-1. Epub 2010 Sep 28. PMID 20878175